# Official Title of Study: -

# MASSAGE WITH SENNA-BASED LAXATIVES VERSUS SENNA-BASED LAXATIVES IN MANAGING OVERFLOW RETENTIVE STOOL INCONTINENCE IN PEDIATRICS: A Randomized Controlled Trial

**Document Date: - 02/12/2020.** 

**Human Subjects protection review board approval** date: - 03/31/2019

# MASSAGE WITH SENNA-BASED LAXATIVES VERSUS SENNA-BASED LAXATIVES IN MANAGING OVERFLOW RETENTIVE STOOL INCONTINENCE IN PEDIATRICS: A

#### **Randomized Controlled Trial**

Nezar Abd Elrouf Abo Halawa

Assistant Lecturer of pediatric surgery, faculty of medicine, South Valley University, Qena, Egypt

Nehad Ahmed youness Abo-Zaid.

Lecture of physical therapy. Department of Physical Therapy for Pediatrics, Faculty of Physical Therapy, South Valley University, Qena, Egypt

#### Abstract

Background: Overflow retentive stool incontinence is a common disorder affecting children that affect the quality of life in the form of shame, humiliation, depression, and decrease reduced self-esteem of children. Aim: To compare the effect of massage with senna-based laxatives versus senna-based laxatives in managing overflow retentive stool incontinence in pediatrics. Methods: Eighty-six children with overflow retentive stool incontinence enrolled in this study and were assessed for eligibility. Children's age ranged from four and fourteen. They were assigned randomly into two groups. Group (A) received abdominal massage with senna-based laxatives and group (B) received senna-based laxatives only. The application of massage was applied for 15 minutes, three times/day for six successive months. Results: Posttreatment there was a significant improvement in both groups in favor of massage group, P < 0.05. Conclusion: Abdominal massage with sennabased laxatives has a great effect on children with overflow retentive stool incontinence than senna-based laxatives only. **Keywords**: Overflow retentive stool incontinence, senna-based laxatives, and abdominal massage.

#### **Introduction**

Constipation is the most common colonic motility disorder in children affecting between 0.7% to 29.6 % of the pediatric population (Rasquin 2006, Mugie 2011) and is frequently associated with fecal incontinence secondary to overflow (Voskuijl 2004)

Laxatives are the main line of maintenance therapy of overflow retentive stool incontinence (ORSI) with satisfying results (Yik 2012) stimulant laxatives like senna based laxatives (SBL) are our standard choice in Egypt due to its availability (Bassiuony 2015).

Massage is the manipulation of muscles and connective tissues (CT) (superficial and deeper layers) by using different techniques. It has been practiced in many ancient civilizations for thousands of years. (Weerapong 2005)

Abdominal massage is a noninvasive, effective, and safe form of constipation management in the general population. (Lamas et al. 2009, Lamas et al., 2012 and Turan&Asti 2016) .It provides a low burden of risk, reduces symptoms of chronic constipation, improves the quality of life, decreases the use of laxatives and increases the frequency and consistency of bowel movements (Smith and Moss, 2008; Moss et al., 2007; Richards 1998; Lamas et al., 2010).

# Subjects and methods:

This randomized controlled study was conducted in the out-patient clinic in the Faculty of Medicine, South Valley University from March 2016 to March 2019. The parents of each child submitted Informed consent. The procedures that followed had No: P.T. REC/012/002277 that approved by the Institutional Ethical Committee Clearance of the Faculty of Physical Therapy at Cairo University. The study had registration number NCT registered on Clinicaltrial.gov.

A total of one hundred and seventy children with overflow retentive stool incontinence were evaluated for eligibility. Twenty-seven children did not complete the treatment course, fifty-eight child excluded due to unresponsiveness or non-compliance to our protocol, and eighty-six child was divided randomly into two groups.

The children were selected according to these criteria: (i) Children's aged ranged from four to fourteen years, (ii) children were from both sexes, (iii) children had a history of overflow retentive stool incontinence. Other children were excluded from our study as they met one of the following criteria:(i) children had suspicion of Hirschsprung's disease, (ii)children had anorectal malformation, (iii) children had organic obstruction, (iv)children failed to complete treatment (if cramping abdominal pain or vomiting occurred), (v) children required bowel surgery.

# Group A: Senna based laxative

Initial cleanout protocol for dis-impaction of the colon with of the administration of one or two enemas per day with 20 ccs/Kg warm tap water with a salt enema (0.9 % saline can be made by adding 1.5 teaspoons of salt to 960 ml of water) (**Levitt 2010**)till been clean by radiologically. If initial dis-impaction was failed or not tolerated, shift to dis-impaction under general anesthesia.

Single 10 mg dose senna was given with the start of impaction. After disimpaction; senna dose was increased if needed by 10 mg/clinic visit/week till achieving no soiling; Documentation of both initial effective starting dose and the time slipped till no soiling. Follow-up visits every month unless soiling recurs if soiling happens; additional dose (by 10 mg) was done. Treatment was continued for 6 months.

At the end of 6 months, the effective ending dose (maintenance dose) was documented.

# Group B: Senna based laxative with massage

Laxative treatment as group A in addition to massage technique.

The massage technique was based upon the Tactile Stimulation Method of Birkestad that primarily consists of palm-to-skin stroking, gentle pressure and static touch (Birkestad 1999).

The patients lying in a comfortable relaxed supine position and physiotherapist performed slow circular clockwise movements on the abdomen, throw tangential pushing, with digital pulp, slow and gradual pressure, with fingers inclination 45

degrees (Harrington & Haskvitz 2006). The pressure applied to the abdomen on each point for 1 min, beginning with the ascending colon, transverse colon, descending colon and sigmoid; this sequence was repeated approximately 15 min. The therapist teaches the parents this technique and asked them to apply at home 3 times/day for 15 min.

# Statistical analysis

The statistical analysis was conducted by using statistical SPSS Package program version 25 for Windows (SPSS, Inc., Chicago, IL). Data were normally distributed by using the Shapiro-Wilk test (parametric data). Additionally, testing for the homogeneity of variance revealed that there was no significant difference (P>0.05). Quantitative descriptive statistics included the mean and standard deviation for demographic data (age, weight, height, and BMI), constipation starting dose, constipation end dose, and time till not soiling variables. Qualitative descriptive statistics included number (percentage) for gender, area, breastfeeding, previous incomplete therapy for constipation, full urinary continence, fissure, psychosocial problems, developmental delay, and history of delayed passage of meconium variables. Using paired t-test to compare between rural area and the urban area within massage group and without massage group for constipation starting dose, constipation end dose, and time till not soiling variables. Using independent t-test to compare between massage group and without massage group for demographic data (age, weight, height, and BMI), constipation starting dose, constipation end dose, and time till not soiling variables. Also, to compare between two groups (massage group and without massage group) within the rural area and urban area for constipation starting dose, constipation end dose, and time till not soiling variables. Chi-square test used to compare between massage group and without the massage group for qualitative variables. All statistical analyses were significant at the level of probability ( $P \le 0.05$ ).

# References:

Rasquin A1, Di Lorenzo C, Forbes D, Guiraldes E, Hyams JS, Staiano A, Walker LS. Gastroenterology. 2006 Apr;130(5):1527-37.

Mugie, S. M., Benninga, M. A., & Di Lorenzo, C. (2011). Epidemiology of constipation in children and adults: A systematic review. Best Practice & Research. Clinical Gastroenterology, 25,3-18.

**Voskuijl WP, Heijmans J, Heijmans HS, Taminiau JA, et al.** Use of Rome II criteria in childhood defecation disorders: applicability in clinical and research practice. J Pediatr 2004;145(2):213–7

Yik YI, Leong LCY, Hutson JM, Southwell BR (2012) The impact of transcutaneous electrical stimulation therapy on appendicectomy operation rates for children with chronic constipation- a single institution experience. J Pediatr Surg47:1421–1426

Ahmed Bassiuony Radwan, Mohammed Soliman El-Debeiky Sameh Abdel-Hay: Contrast enema as a guide for senna-based laxatives in managing overflow retentive stool incontinence in pediatrics PediatrSurgInt (2015) 31:765–771

**Levitt MA, Pen~aA:**(2010) Fecal incontinence and constipation. In: Holcomb GW III, Murphy JP (eds) Ashcraft's pediatric surgery, 5th ed. Saunders Elsevier, Philadelphia, pp 491–501

Suzanne M. Mugie, Carlo Di Lorenzo & Benninga. Constipation in childhood. Nature Volume 8, pages 502–511 (2011)

Voskuijl W, de Lorijn F, Verwijs W, Hogeman P, Heijmans J, Makel M, et al. PEG 3350 (Transipeg) versus lactulose in the treatment of childhood functional constipation: a double-blind, randomized, controlled, multicentre trial. Gut 2004;53:1590–4.

Nurko S, Youssef NN, Sabri M, Langseder A, McGowan J, Cleveland M, et al. PEG3350 in the treatment of childhood constipation: a multicentre, double-blinded, placebo-controlled trial. J Pediatr 2008;153(2):254–61. 261 e1

**Bischoff A, Brisighelli G, Dickie B, Frischer J, Levitt MA&Peña A**. Idiopathic constipation: A challenging but manageable problem. J Pediatr Surg. 2018 Sep;53(9):1742-1747.

Clarke MC, Chase JW, Gibb S, et al. Decreased colonic transit time after transcutaneous interferential electrical stimulation in children with slow-transit constipation. J PediatrSurg 2009;44:408–12

**RajindrajithS, Devanarayana NM.** Constipation in children: novel insight into epidemiology, pathophysiology, and management. J NeurogastroenterolMotil 2011;17: 35–47.

**Brazzell M, Griffiths P.**Behavioural and cognitive interventions with or without other treatments for the management of fecal incontinence in children. Cochrane Database Syst Rev 2006;2: CD002240. https://doi.org/10.1002/14651858.CD002240.pub3.

Yik YI, Ismail KA, Hutson JM, et al. Home transcutaneous electrical stimulation to treat children with slow-transit constipation. J PediatrSurg 2012;47:1285–90

**Tabbers MM, DiLorenzo C, Berger MY et al** (2014) Evaluation and treatment of functional constipation in infants and children: evidence-based recommendations from ESPGHAN and NASPGHAN. J PediatrGastroenterolNutr 58(2):258–274

Ayas S<sub>2</sub>, Leblebici B., Sozay. S, Bayramo glu M. and. Niron E. A.: "The effect of abdominal massage on bowel function in patients with spinal cord injury," American Journal of Physical Medicine and Rehabilitation, vol. 85, no. 12, pp. 951–955, 2006.

**Benninga MA, Voskuijl WP, Taminiau JAJ.** Childhood constipation: is there new light in the tunnel? J PediatrGastroenterolNutr 2004; 39: 448–64.CrossrefCASPubMedWeb of Science®Google Scholar

**Bharucha AE.:** Lower gastrointestinal functions. NeurogastroenterolMotil 2008; 20: 103–13. Wiley Online LibraryPubMedWeb of Science®Google Scholar

- **Bromley D.:** "Abdominal massage in the management of chronic constipation for children with disability," Community Practitioner, vol. 87, no. 12, pp. 25–29, 2014.
- **Diego MA et al** (2007) Preterm infant massage elicits consistent increases in vagal activity and gastric motility that are associated with greater weight gain. ActaPaediatrica; 96: 11, 1588–1591.
- **Emly M.:** "Abdominal massage for adults with learning disabilities" Nursing Times, vol. 97, no. 30, pp. 61–62, 2001.
- *Harrington KL, Haskvitz EM.* Managing patient's constipation with physical therapy. PhysTher 2006; 86 1511–9.
- Lämäs K, Lindholm L, Engström B, Jacobsson C. Abdominal massage for people with constipation: a cost-utility analysis. J AdvNurs 2010; 66: 1719–29.
- **Lämäs K., Graneheim U. H., and Jacobsson C.:** "Experiences of abdominal massage for constipation," Journal of Clinical Nursing, vol. 21, no. 5-6, pp. 757–765, 2012.
- Lämäs K., Lindholm L., Stenlund H., Engstrom B., and Jacobsson C.: "Effects of abdominal massage in the management of constipation: a randomized controlled trial," International Journal of Nursing Studies, vol. 46, no. 6, pp. 759–767, 2009.
- Liu Z., Sakakibara R., Odaka T.et al.: Mechanism of abdominal massage for difficult defecation in a patient with myelopathy (HAM/TSP)," Journal of Neurology, vol. 252, no. 10, pp. 1280–1282, 2005.
- **McClurg D, Lowe-Strong A.** Does abdominal massage relieve constipation? Nurs Times 2011; 107: 20–2.PubMedGoogle Scholar
- Moss L., Smith M., Wharton S., and Hames A.: "Abdominal massage for the treatment of idiopathic constipation in children with profound learning disabilities: a single case study design," British Journal of Learning Disabilities, vol. 36, no. 2, pp. 102–108, 2008.

- Nam MJ, Bang Y, Kim TI.: Effects of abdominal meridian massage with aroma oils on relief of constipation among hospitalized children with brain-related disabilities. J Korean AcadNurs. 2013; 43: 247–255.
- **Preece J.:** "Introducing abdominal massage in palliative care for the relief of constipation," Complementary Therapies in Nursing and Midwifery, vol. 8, no. 2, pp. 101–105, 2002.
- **Turan N. and. Asti T. A:** "The effect of abdominal massage on constipation and quality of life," Gastroenterology Nursing, vol. 39, no. 1, pp. 48–59, 2016.
- **Turnbull GK, Lennard-Jones JE, Bartram CI.** (1986) Failure of rectal expulsion as a cause of constipation: why fiber and laxatives sometimes fail. Lancet1(8484): 767–9
- Weerapong P., Hume P. A., and Kolt G. S.: "The mechanisms of massage and effects on performance, muscle recovery and injury prevention," Sports Medicine, vol. 35, no. 3, pp. 235–256, 2005.
- **Le Blanc-Louvry I., et al.:** Feb 2002. Does mechanical massage of the abdominal wall after colectomy reduce post-operative pain and shorten the duration of ileus: results of a randomized study. Journal of Gastrointestinal Surgery 6 (1), 43e49.
- **Faleiros FT, Machado NC:** Assessment of health-related quality of life in children with functional defecation disorders. J Pediatr (Rio J) 2006;82:421–425.